CLINICAL TRIAL: NCT05525546
Title: Phase 1 Randomized, Placebo-Controlled, Study to Compare the Safety, Reactogenicity, and Immunogenicity of a Full-Strength Formulation of Trivalent Salmonella (S. Enteritidis/S. Typhimurium/S. Typhi Vi) Conjugate Vaccine (TSCV), a Half-Strength Formulation of TSCV, and a Dilutional Half-Strength Dose of TSCV Against Invasive Salmonella Disease Administered Parenterally to Healthy U.S. Adults
Brief Title: Salmonella Conjugates CVD 2000: Study of Responses to Vaccination With Trivalent Salmonella Conjugate Vaccine to Prevent Invasive Salmonella Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Wilbur Chen, MD, MS, Professor of Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HP-00099225
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Risk Reduction
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A: Full-Strength Formulation (Experimental): Individuals receive one dose of full-strength Trivalent Salmonella Conjugate Vaccine (TSCV). Subsequent blood samples are taken for safety and immunological testing.
  Interventions: Biological: Trivalent Salmonella Conjugate Vaccine (TSCV) Full-Strength Formulation
- Group B: Half-Strength Formulation (Experimental): Individuals receive one dose of half-strength Trivalent Salmonella Conjugate Vaccine (TSCV). Subsequent blood samples are taken for safety and immunological testing.
  Interventions: Biological: Trivalent Salmonella Conjugate Vaccine (TSCV) Half-Strength Formulation
- Group C: Dilutional Half-Strength Formulation (Experimental): Individuals receive one dose of dilutional half-strength Trivalent Salmonella Conjugate Vaccine (TSCV). Subsequent blood samples are taken for safety and immunological testing.
  Interventions: Biological: Trivalent Salmonella Conjugate Vaccine (TSCV) Dilutional Half-Strength Formulation
- Group D: Placebo (Placebo Comparator): Individuals receive one dose of placebo. Subsequent blood samples are taken for safety and immunological testing.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Trivalent Salmonella Conjugate Vaccine (TSCV) Full-Strength Formulation — One dose of the full-strength conjugate vaccine is administered via an intramuscular injection in to the deltoid muscle on Study Day 1. The full-strength conjugate vaccine consists of 25 mcg of each conjugate; Salmonella Enteritidis, Salmonella Typhimurium, and Salmonella Typhi Vi.
  Arms: Group A: Full-Strength Formulation
Biological: Trivalent Salmonella Conjugate Vaccine (TSCV) Half-Strength Formulation — One dose of the half-strength conjugate vaccine is administered via an intramuscular injection in to the deltoid muscle on Study Day 1. The half-strength conjugate vaccine consists of 12.5 mcg of Salmonella Enteritidis, 12.5 mg of Salmonella Typhimurium, and 25 mcg of Salmonella Typhi Vi.
  Arms: Group B: Half-Strength Formulation
Biological: Trivalent Salmonella Conjugate Vaccine (TSCV) Dilutional Half-Strength Formulation — One dose of the dilutional half-strength conjugate vaccine is administered via an intramuscular injection in to the deltoid muscle on Study Day 1. The dilutional half-strength conjugate vaccine consists of 12.5 mcg of each conjugate; Salmonella Enteritidis, Salmonella Typhimurium, and Salmonella Typhi Vi.
  Arms: Group C: Dilutional Half-Strength Formulation
Other: Placebo — One dose of placebo is administered via an intramuscular injection in to the deltoid muscle on Study Day 1. The placebo consists of sterile phosphate-buffered saline (PBS) solution containing polysorbate 80, and 2-phenoxyethanol preservative.
  Arms: Group D: Placebo

SUMMARY:
This is a randomized, placebo-controlled interventional study. The main purpose of this research is to test the safety and measure the immune response of the trivalent vaccine against invasive Salmonella disease. The vaccine will be tested over a range of doses.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Age 18 - 49 years, inclusive
* Good general health as determined by: vital signs (heart rate <100 bpm; blood pressure systolic >90 mm Hg and ≤150 mm Hg; diastolic >45 mm Hg and ≤90 mm Hg; oral temperature <100.4ºF), medical history, and a physical examination† within 45 days before administration of first dose of vaccine.

  † The intent is to evaluate for acute or ongoing chronic medical conditions which have been present for 90 days or more and which could affect the assess of safety or immunogenicity. Chronic medical conditions should be stable for at least 60 days; defined as no hospitalizations, ER, or urgent care for medical intervention and no change in chronic prescription medications for at least 60 days. Changes in medications due to insurance or financial reasons and when within the same class of medications or changes for improvements in medical conditions are not exclusionary. Medications which are taken prn are also no exclusionary.
* Expressed interest and availability to fulfill the study requirements
* For females of child-bearing potential*, must agree to acceptable birth control &, 4 weeks before enrollment and through 4 weeks after last vaccination.

  * females of child-bearing potential are defined as: not sterilized via tubal ligation, bilateral oophorectomy, salpingectomy, hysterectomy, or successful Essure® placement (permanent, nonsurgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or <1 year of the last menses if menopausal.

  & acceptable birth control includes: non-male sexual relationships, abstinence from sexual intercourse with a male partner, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more prior to the subject receiving the first study vaccination, barrier methods such as condoms or diaphragms with spermicide or foam, effective intrauterine devices, NuvaRing®, and licensed hormonal methods such as implants, injectables, or oral contraceptives.
* Agrees not to participate in another clinical trial at any time during the study period.
* Agrees to allow for the indefinite storage of blood samples for future research use.
* Complies with Pharmaron's Coronavirus disease 2019 (Covid 19) policy.

Exclusion Criteria:

* History of typhoid vaccination or known history of typhoid infection within 5 years
* Unacceptable laboratory abnormality from screening (prior to first vaccination) or upon safety laboratory testing (prior to second vaccination) as listed below. Laboratories with abnormalities which are possibly transient in nature may be repeated one time.

  1. Hemoglobin, white blood cell (WBC) count, absolute neutrophil count (ANC), or platelet count of an unacceptable value
  2. Creatinine, Aspartate Aminotransferase (AST), Alanine aminotransferase (ALT), total bilirubin, or C-reactive protein of an unacceptable value c. Positive serology for hepatitis C or HIV antibody or hepatitis B surface antigen.

(Subjects will be informed if their results are positive for hepatitis C, Human Immunodeficiency Virus (HIV) antibody or hepatitis B surface antigen and will be referred to a primary care provider for follow up of these abnormal laboratory tests.)

* For women of child-bearing potential, positive serum pregnancy test (during screening within 45 days of enrollment) or positive urine pregnancy test (prior to and within 24 hours of administering each dose of vaccine).
* Nursing mother.
* Temperature > 38.0°C (100.4°F) or symptoms of an acute self-limited illness such as an upper respiratory infection or gastroenteritis within 3 days prior to vaccination.
* This exclusion criterion is to be used for the duration that there is a U.S. Public Health Emergency for COVID-19; once the declaration has ended, this criterion will not be used. Temperature > 38.0°C (100.4°F) or symptoms of a COVID-19 infection# within 10 days prior to vaccination.

  * Symptoms of a COVID-19 infection include fever, chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, and diarrhea.

https://www.cdc.gov/coronavirus/2019-ncov/symptoms-testing/symptoms.html

* Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* Diagnosis of schizophrenia or other major psychiatric disease
* Failure to pass the Comprehension Assessment Tool test during screening (70% correct answers are required to pass. Subjects will be provided the opportunity to repeat the test once).
* Receipt of an experimental agent (vaccine, drug, device, etc.) within 28 days before enrollment or expects to receive an experimental agent during the study period.
* Receipt of any licensed vaccine within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) before enrollment in this study.
* Known sensitivity to any ingredient in the study vaccine, including a history of severe allergic reaction to tetanus vaccine.
* Receipt of immunoglobulin or other blood product within the 3 months prior to vaccination in this study.
* Immunosuppression as a result of an underlying illness or treatment with immunosuppressive or cytotoxic drugs, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months.
* Long-term use (>2 weeks) of oral or parenteral steroids (glucocorticoids), or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (nasal and topical steroids are allowed).
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
Frequency and Severity of Solicited Local and Systemic Adverse Events (AEs) | Approximately six months
  To assess the frequency and severity of solicited local (i.e., injective site) and systemic (such as fever) AEs during the first 7 days following each dose of vaccine.
Frequency and Severity of Unsolicited AEs and Serious Adverse Events (SAEs) | Approximately six months
  To assess the frequency and severity of unsolicited AEs within 28 days of each dose of vaccine and the occurrence of any SAEs through 6 months after the last dose of vaccine
Proportion of Responders | approximately six months
  To measure the proportion of subjects that achieve a four-fold increase in titer, as compared to baseline, of specific serum Immunoglobulin G (IgG) anti-Core-O polysaccharide (anti-COPS) (S. Enteritidis or S. Typhimurium), anti-Vi (S. Typhi) polysaccharide, and anti-Flagellin subunit protein (anti-FliC) (S. Enteritidis or S. Typhimurium) antibody at day 29, as measured by Enzyme-linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Myron M Levine, MD, DTPH, Study Director — University of Maryland, Baltimore
Locations (1):
- Pharmaron, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No